CLINICAL TRIAL: NCT05439317
Title: Elasticity of the Hoffa's Fat Pad in Patients With Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-09-013AC
Record Dates: First submitted 2022-05-19; First posted 2022-06-30 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Knee Osteoarthritis; Elasticity Imaging Techniques
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- knee osteoarthritis group: individuals being diagnosed with osteoarthritis and classified by K-L grading
- healthy group: individuals without knee pain or diagnosis of knee osteoarthritis

SUMMARY:
Knee osteoarthritis (OA) is a common problem in clinical settings. Knee OA is well known for its association with the wear and tear of the cartilage and osteophyte formation. Evidence has suggested the importance of the infrapatellar fat pad, known as Hoffa's fat pad, during the development of knee OA. Some studies have demonstrated the protective role of the infrapatellar fat pad, whereas others have suggested an inflammatory role such as increased fibrosis and proinflammatory cytokine levels. Ultrasound is exceptionally convenient in the assessment of the musculoskeletal system, and elastography is a tool to evaluate tissue texture. Therefore, in this study, we investigated the Hoffa's fat pad in knee OA patients by using elastography.

DETAILED DESCRIPTION:
This was an observation study that included a control group. We enrolled 20 patients with knee OA, as well as 10 healthy individuals. The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and Kellgren-Lawrence X-ray grading were employed to determine disease severity. All the study participants received elastography assessment, including strain and shear wave elastography in the knee extension and flexion position. The strain elastography contained color mapping that enabled the calculation of the relative texture and strain ratio. The shear wave elastography revealed the qualitative velocity, which was measured 3 times. Each patients with knee OA received elastography examination twice: once before hyaluronic acid injection and once 1 month after the injection.

ELIGIBILITY:
Inclusion Criteria:

OA group

* Kellgren-Lawrence grading I-IV proved by knee X-ray Healthy group
* No knee pain or received injection during the past 1 year
* No history of knee OA

Exclusion Criteria:

* History of knee surgery, trauma or malignancy
* History of patellar tendinopathy or patellofemoral pain syndrome
* Refused informed consent

Ages: 20 Years to 86 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: individuals with knee osteoarthritis diagnosis is classified as K-L grading I - IV individuals in control group has no knee pain or osteoarthritis history
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
shear modulus | before and 1-3 months after hyaluronic acid injection
  the absolute quantitative measurement of elasticity (kPa) of Hoffa's fat pad
strain ratio | before and 1-3 months after hyaluronic acid injection
  the semiquantitative measurement of elasticity of Hoffa's fat pad, a ratio with patellar tendon as reference
thickness of Hoffa's fat pad | before and 1-3 months after hyaluronic acid injection
  the thickness of Hoffa's fat pad from mid patellar tendon to femur cartilage

CONTACTS AND LOCATIONS:
Overall Officials: Ding-Hao Liu, Study Chair — Physical and Rehabilitation Medicine, Veterans General Hospital
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan